CLINICAL TRIAL: NCT04304040
Title: A Phase I/IIa Study on Dose-escalation and Extension of Recombinant Humanized Type II CD20 Monoclonal Antibody MIL62 Injection Combined With BTK Inhibitor Orelabrutinib in the Treatment of Recurrent/Refractory CD20+B-cell Lymphoma
Brief Title: A Study of MIL62 Combined With Orelabrutinib for the Treatment of R/R CD20+B Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIL62-CT03
Record Dates: First submitted 2020-03-05; First posted 2020-03-11 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: B-cell Lymphoma Recurrent; B-cell Lymphoma Refractory
Keywords: CD20+
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Orelabrutinib; Drug: Recombinant humanized monoclonal antibody MIL62 injection

INTERVENTIONS:
Drug: Orelabrutinib — BTK inhibitor Orelabrutinib low dose or high dose; Part A:28days/cycle, Cycle1:35days; Part B:21 days/cycle, Cycle1:28days.
Drug: Recombinant humanized monoclonal antibody MIL62 injection — Recombinant humanized monoclonal antibody MIL62 injection, 800mg or1000mg each time, Part A:28days/cycle, Cycle1:35days; Part B:21 days/cycle, Cycle1:28days.

SUMMARY:
Dose escalation and expansion phase I/IIa clinical study of recombinant humanized type II CD20 monoclonal antibody MIL62 injection combined with a novel selective Bruton Tyrosine Kinase(BTK) inhibitor Orelabrutinib in the treatment of recurrent/refractory CD20+B cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, gender not limited
2. Dose escalation phase: Histologically confirmed CD20 positive B-cell non-Hodgkin's lymphoma; Expansion stage: R/R NHL Or histologically diagnosed CD20 positive chronic lymphocytic leukemia/small lymphocytic lymphoma;
3. Dose escalation phase ：Patients who have received at least one treatment regimen Expansion stage：Patients who have received at least one to four treatment regimens with at least one regimen containing rituximab;
4. Eastern cancer collaboration group(ECOG) physical status score: 0-2
5. Laboratory tests performed within 7 days prior to the first acceptance of the study drug met the protocol criteria.
6. Expected survival ≥6 months
7. Sign a written informed consent.

Exclusion Criteria:

1. Expansion stage: DLBCL transformed from follicular lymphoma, DLBCL with follicular lymphoma, and lymphomas with primary or central nervous system involvement.
2. Received any of the anti-tumor treatments(note in the protocol) before the first study drug.
3. Previous use of any anticancer vaccine.
4. Patients who had received hematopoietic stem cell transplantation within 3 months before the first administration
5. Patients scheduled for major surgery within 28 days prior to initial administration or during the expected study period.
6. Patients who Is participating in other clinical trials or first administration less than 28 days after the end of the previous clinical trial.
7. Receiving prednisone treatment or other corticosteroid treatment with the same dose as prednisone ;Patients who require warfarin or an equivalent vitamin K antagonist;
8. During the study period, drugs with moderate or severe inhibition or strong induction of cytochrome CYP3A4 were taken together;
9. Subject has a history of any of the diseases note in the protocol;
10. Patients with infections;
11. Impact testing scheme compliance or other serious results explain the poor control of the merger of the disease(note in the protocol);
12. Toxicity of any previous anticancer treatment has not recovered to ≤1, except for hair loss;
13. A history of severe allergic reactions to humanized monoclonal antibodies or known allergies to any component of Orelabrutinib or MIL62;
14. Inability to swallow research drugs, or the presence of conditions that significantly affect gastrointestinal function;
15. Hepatitis b surface antigen (HBsAg) and/or hepatitis b core antibody (HBcAb) are positive ; Hepatitis c virus (HCV) antibody positive and HCV RNA positive patients; Human immunodeficiency virus (HIV) serum response was positive;
16. Pregnant and lactating women; For women of childbearing age who have not undergone sterilization surgery: do not agree to use appropriate methods of contraception;
17. For men not undergoing sterilization: do not agree to use the barrier method of contraception;
18. Other circumstances considered inappropriate for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT)(Dose escalation phase) | At the end of Cycle 1 (each cycle is 28 days)
  Safety observation indicator
Maximum tolerated dose (MTD) (Dose escalation phase) | At the end of Cycle 1 (each cycle is 28 days)
  Safety observation indicator
Recommended dose for phase 2 trials of two-drug combinations (RP2D) (Dose escalation phase) | At the end of Cycle 1 (each cycle is 28 days)
  Safety observation indicator
objective remission rate(ORR) (Dose expansion phase) | At the end of Cycle 30 (each cycle is 28 days)
  Efficacy observation indicator

SECONDARY OUTCOMES:
objective remission rate(ORR) | At the end of Cycle 30 (each cycle is 28 days)
  Efficacy observation indicator
Area under the plasma concentration vs time curve(AUC) | At the end of Cycle 6 (each cycle is 28 days)
  pharmacokinetic parameter of MIL62 combined with Orelabrutinib in the treatment
Apparent half-life for designated elimination phases (t½) | At the end of Cycle 6 (each cycle is 28 days)
  pharmacokinetic parameter of MIL62 combined with Orelabrutinib in the treatment
The peak plasma concentration (Cmax) | At the end of Cycle 6 (each cycle is 28 days)
  pharmacokinetic parameter of MIL62 combined with Orelabrutinib in the treatment
Duration of remission(DOR) | 3 years after first treatment
  Efficacy observation indicator
Progression-free survival(PFS) in the treatment of R/R CD20+B cell lymphoma | 3 years after first treatment
  Preliminary evaluation of MIL62 combined with Orelabrutinib in the treatment of relapsed/refractory CD20+B cell lymphoma with 3-year progression-free survival
overall survival(OS) in the treatment of R/R CD20+B cell lymphoma | 3 years after first treatment
  Preliminary evaluation of MIL62 combined with Orelabrutinib in the treatment of recurrent/refractory CD20+B cell lymphoma with 3-year overall survival
Duration of remission(DOR) in the treatment of R/R NHL | 3 years after first treatment
  Preliminary evaluation of remission duration of MIL62 combined with Orelabrutinib in the treatment of Recurrent/refractory Non Hodgkin Lymphoma
Progression-free survival(PFS) in the treatment of R/R NHL | 3 years after first treatment
  Preliminary evaluation of MIL62 combined with Orelabrutinib in the treatment of Recurrent/refractory Non Hodgkin Lymphoma with 3-year progression-free survival
overall survival(OS) in the treatment of R/R NHL | 3 years after first treatment
  Preliminary evaluation of MIL62 combined with Orelabrutinib in the treatment of Recurrent/refractory Non Hodgkin Lymphoma with 3-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (10):
- China (10):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan hospital, capital medical university, Beijing, Beijing Municipality
  - Cancer hospital, Chinese academy of medical sciences, Beijing, Beijing Municipality
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No